CLINICAL TRIAL: NCT07272785
Title: Maternal Informing on Labor Induction: Impact on Childbirth Experience
Status: Recruiting | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: OP2025/8882
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-11

CONDITIONS: Labor, Induced; Labor, Obstetric; Pregnancy; Humans; Prospective Study; Prospective Study , Questionaires; Childbirth Experience
Keywords: Childbirth experience; Induction of labor; Pregnancy; Childbirth; Obstetrics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subject undergoing planned induction of labor

SUMMARY:
The aim of this study is to explore the information provided to mothers about labor induction and its connection to their childbirth experience. In addition, the study examines how the use of social media may influence the birth experience among patients undergoing labor induction.

DETAILED DESCRIPTION:
Subject undergoing planned induction of labor will be recruited. At recruitment the participants will be asked to answer a questionnaire. Follow-up questionnaires will be sent to the participants one week and three months after the induction.

The first questionnaire assesses how well the participants were informed about the induction. The following questionnaires will assess the childbirth experience and induction experience.

The main aim of the study is to investigate whether being being well informed about the induction of labor is related to better experience of childbirth. Moreover, the correlation between reported social media use and childbirth experience will be evaluated.

After obtaining full data from the first 50 subjects an interim analysis will be performed, to decide the final target sample size.

ELIGIBILITY:
Inclusion Criteria:

* Planned induction of labor at the antenatal ward or at the outpatient clinic
* Adequate language skills (Finnish, Swedish, English)

Exclusion Criteria:

* Induction at the delivery ward or at the obstetric emergency care clinic
* Spontaneous onset of labor or a planned cesarean delivery
* Age below 18 years at the time of recruitment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant subjects undergoing planned induction for various reasons.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Childbirth experience | Three months after induction of labor
  Childbirth experience assessed using visual analog scale (VAS) where 0 is the worst possible and 10 the best possible childbirth experience.

SECONDARY OUTCOMES:
Childbirth experience | One week after induction of labor
  Childbirth experience assessed using visual analog scale (VAS) where 0 is the worst possible and 10 the best possible childbirth experience.
Experience of labor induction | One week after induction of labor
  Assessed using visual analog scale (VAS) where 0 is the worst possible and 10 the best possible labor induction experience.
Experience of labor induction | Three months after induction of labor
  Assessed using visual analog scale (VAS) where 0 is the worst possible and 10 the best possible labor induction experience.
Did childbirth experience meet participant's expectations | One week after induction of labor
  Four points Likert scale with the following possible answers: 1) very poorly, 2) quite poorly, 3) quite well, 4) very well.

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Huhtala, M.D., Ph.D., Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: No
To ensure study subject anonymity the study data will not be published.